CLINICAL TRIAL: NCT03272373
Title: NexGen® TM Tibia Clinical Outcomes Study: Prospective Multicenter Study of the NexGen® TM Monoblock and Modular Tibias
Brief Title: NexGen TM Tibia Clinical Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K.CR.I.G.16.34
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Polyarthritis; Collagen Disorders and/or Avascular Necrosis of the Femoral Condyle; Post-traumatic Loss of Joint Configuration; Moderate Valgus, Varus, or Flexion Deformities
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Intervention Model Description: 2 single arms being analyzed separately
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Monoblock (Other): Subjects that receive the NexGen TM Monoblock Tibia
  Interventions: Device: NexGen TM Monoblock Tibia
- Modular (Other): Subjects that receive the NexGen TM Modular Tibia
  Interventions: Device: NexGen TM Modular Tibia

INTERVENTIONS:
Device: NexGen TM Monoblock Tibia — Primary cementless tibia total knee arthroplasty
  Arms: Monoblock
Device: NexGen TM Modular Tibia — Primary cementless tibia total knee arthroplasty
  Arms: Modular

SUMMARY:
The objective of this study is to evaluate clinical performance for the commercially available NexGen TM Monoblock Tibia and NexGen TM Modular Tibia used in primary cementless tibia total knee arthroplasty.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized clinical study designed to facilitate the collection and evaluation of radiographic parameters, pain and function, survival of the device, and adverse event data. This clinical study will include the NexGen TM Monoblock Tibia and NexGen TM Modular Tibia as 2 single-arms being analyzed separately.

The study will require each site to obtain IRB approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their cementless tibia total knee arthroplasty. An immediate postoperative radiograph will be required. Postoperative clinical follow-up and radiographic evaluations will be conducted at 6 weeks, 6 months, 1 year, and 2 years.

The primary endpoint of this study is to evaluate the clinical performance of the implant at 2 years postoperatively using radiographic parameters. Radiographs will be assessed for the absence of progressive tibial radiolucencies, as defined in the radiographic protocol.

The secondary endpoints of this study will evaluate the clinical performance of the implant at 2 years postoperatively, based upon:

* No revisions for any reason
* Oxford Knee Score >38

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age.
2. Patient qualifies for a primary cementless tibia total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

   1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis.
   2. Collagen disorders and/or avascular necrosis of the femoral condyle.
   3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy.
   4. Moderate valgus, varus, or flexion deformities.
   5. The salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee.
3. Patient has participated in the study-related Informed Consent process.
4. Patient is willing and able to provide written Informed Consent by signing and dating the IRB approved Informed Consent Form.
5. Patient is willing and able to complete scheduled study procedures and follow-up evaluations as described in the Informed Consent Form.
6. Independent of study participation, patient is a candidate for commercially available cementless NexGen TM tibial knee component, implanted in accordance with product labeling.

Exclusion Criteria:

1. Previous history of infection in the affected joint.
2. Active local or systemic infection that may affect the prosthetic joint.
3. Insufficient bone stock on femoral or tibial surfaces.
4. Skeletal immaturity.
5. Neuropathic arthropathy.
6. Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb.
7. A stable, painless arthrodesis in a satisfactory functional position.
8. Severe instability secondary to the absence of collateral ligament integrity.
9. Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin.
10. Patient has previously received partial or total knee arthroplasty for the ipsilateral knee.
11. Patient is currently participating in any other surgical intervention studies or pain management studies.
12. Patient is known to be pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.).
13. Patient has a known or suspected sensitivity or allergy to one or more of the implant materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, RN, MBA, Study Director — Zimmer Biomet
Locations (7):
- United States (7):
  - LA BioMed at Harbor-UCLA Medical Center, Torrance, California
  - Cornerstone Orthopaedics & Sports Medicine, P.C., Wheat Ridge, Colorado
  - Franciscan Health, Mooresville, Indiana
  - Henry County Orthopedics and Sports Medicine, New Castle, Indiana
  - Woods Mill Orthopedics, Ltd, Chesterfield, Missouri
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Knees
Groups:
- NexGen TM Monoblock Tibia: NexGen Trabecular Metal (TM) Monoblock Tibia used in primary cementless total knee arthroplasty
- NexGen TM Modular Tibia: NexGen Trabecular Metal (TM) Modular Tibia used in primary cementless total knee arthroplasty
Period: Overall Study
Arm/Group | NexGen TM Monoblock Tibia | NexGen TM Modular Tibia
Started | 104; 110 Knees (104 participants (110 knees) proceeded with surgery and received the NexGen TM Monoblock Tibia implant (study device). There were 98 participants with surgery on one knee and 6 participants with surgery on both knees.) | 56; 63 Knees (56 participants (63 knees) proceeded with surgery and received the NexGen TM Modular Tibia implant (study device). There were 49 participants with surgery on one knee and 7 participants with surgery on both knees.)
Completed | 83; 89 Knees (83 participants (89 knees) completed the 2 year follow-up physical exam.) | 48; 55 Knees (48 participants (55 knees) completed the 2 year follow-up physical exam.)
Not Completed | 21; 21 Knees | 8; 8 Knees

BASELINE CHARACTERISTICS:
Population: Demographics are being reported for the 110 knees that received the NexGen TM Monoblock Tibia implant and the 63 knees that received the NexGen TM Modular implant (study devices).
Units Other Than Participants: Knees
Groups:
- Total: Total of all reporting groups
Arm/Group | NexGen TM Monoblock Tibia | NexGen TM Modular Tibia | Total
Number analyzed (Participants) | 104 | 56 | 160
Number analyzed (Knees) | 110 | 63 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.60 (7.78) | 61.37 (8.14) | 62.15 (7.91)
Sex: Female, Male [Count of Units; unit: Knees]
  Female | 66 | 36 | 102
  Male | 44 | 27 | 71
Race/Ethnicity, Customized [Count of Units; unit: Knees]
  African American or Black | 9 | 0 | 9
  Asian | 1 | 0 | 1
  Hispanic or Latino | 19 | 4 | 23
  White | 69 | 59 | 128
  Not Recorded | 12 | 0 | 12
Region of Enrollment [Number; unit: Knees]
  United States | 110 | 63 | 173

OUTCOME MEASURES:

1. Primary Outcome: Radiograph Assessment of Progressive Tibial Radiolucencies
Description: Progressive tibial radiolucency will be derived in accordance with the following definitions:
  Absent: No evidence of an increase in either radiolucency extent (number of zones involved) or measured width within a zone.
  Present: Presence of either: An increase in the number of zones with a measured tibial radiolucency, OR an increase in the measured tibial radiolucency width within a zone of >0.5mm.
  Unable to assess: One or more of the component factors necessary to derive progressive tibial radiolucency is unavailable.
Time Frame: 2 years
Population: Monoblock: 77 participants (83 knees) had radiographs analyzed at the 2 year follow-up interval.
  Modular: 48 participants (55 knees) had radiographs analyzed at the 2 year follow-up interval.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | NexGen TM Monoblock Tibia | NexGen TM Modular Tibia
Number analyzed (Participants) | 77 | 48
Number analyzed (Knees) | 83 | 55
Knees
  Absent | 82 | 55
  Present | 0 | 0
  Unable to assess | 1 | 0

2. Secondary Outcome: Oxford Knee Score
Description: The Oxford Knee Score is a patient completed 12 question metric to rate a patient's knee pain and function using an ordinal 0 - 4 point scale. The total score is obtained by calculating the sum of the 12 items. The maximum score is 48 points (best) and the minimum score is 0 points (worst).
Time Frame: 2 years
Population: Monoblock: 83 participants (89 knees) completed the Oxford Knee Score (OKS) at the 2 year interval.
  Modular: 46 participants (52 knees) completed the Oxford Knee Score (OKS) at the 2 year interval.
  Oxford Knee Scores above 41 are considered excellent and scores from 34 to 41 are considered good. The endpoint was designed to distinguish scores above 38. Reference: Murray et al. (2007). The use of the Oxford hip and knee scores. Bone & Joint Journal, 89(8), 1010-1014
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | NexGen TM Monoblock Tibia | NexGen TM Modular Tibia
Number analyzed (Participants) | 83 | 46
Number analyzed (Knees) | 89 | 52
Knees
  OKS >38 | 64 | 47
  OKS <=38 | 25 | 5

3. Secondary Outcome: Revision Rate
Description: Rate of the number of revisions for any reason
Time Frame: 2 years
Population: A revision is when the study implant is removed/revised due to an adverse event. Of the 110 knees that received the NexGen TM Monoblock Tibia implant, there were 2 reported revisions. Of the 63 knees that received the NexGen TM Modular Tibia implant, there were 0 reported revisions
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | NexGen TM Monoblock Tibia | NexGen TM Modular Tibia
Number analyzed (Participants) | 104 | 56
Number analyzed (Knees) | 110 | 63
Knees
  Number of knees not revised | 108 | 63
  Number of knees revised | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the date of study device surgery through the 2 year follow-up interval. An exception is for the participants who did not complete the study, where adverse events were collected through the date of when the participant exited the study.
Arm/Group | NexGen TM Monoblock Tibia | NexGen TM Modular Tibia
All-Cause Mortality (participants affected / at risk) | 2/104 | 0/56
Serious Adverse Events (participants affected / at risk) | 10/104 | 7/56
Other Adverse Events (participants affected / at risk) | 39/104 | 28/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NexGen TM Monoblock Tibia (N=104) | NexGen TM Modular Tibia (N=56)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0) — General adverse event (not study knee)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) — General adverse event (not study knee)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) — General adverse event (not study knee)
Genitourinary/Renal (Renal and urinary disorders) | 1 (1) | 0 (0) — General adverse event (not study knee)
Musculoskeletal (not study knee) (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) — General adverse event (not study knee)
Neurological (Nervous system disorders) | 0 (0) | 1 (1) — General adverse event (not study knee)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — General adverse event (not study knee)
Contralateral Knee Replacement (UKA or TKA) (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) — General adverse event (not study knee)
Traumatic Injury (not study knee) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — General adverse event (not study knee)
Deep Wound Infection (Infections and infestations) | 2 (2) | 0 (0) — Study knee related
Other General Adverse Event (General disorders) | 3 (3) | 0 (0) — General adverse event (not study knee)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NexGen TM Monoblock Tibia (N=104) | NexGen TM Modular Tibia (N=56)
Cardiovascular (Cardiac disorders) | 5 (5) | 0 (0) — General adverse event (not study knee)
Neurological (Nervous system disorders) | 2 (5) | 0 (0) — General adverse event (not study knee)
Oncological (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) — General adverse event (not study knee)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — General adverse event (not study knee)
Contralateral Knee Replacement (UKA or TKA) (Surgical and medical procedures) | 3 (3) | 5 (5) — General adverse event (not study knee)
Vascular/DVT (Vascular disorders) | 3 (3) | 1 (1) — General adverse event (not study knee)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — General adverse event (not study knee)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) — General adverse event (not study knee)
Stiffness/Limited ROM (progressive/persistent) (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) — Study knee related
Genitourinary/Renal (Renal and urinary disorders) | 1 (1) | 0 (0) — General adverse event (not study knee)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Study knee related
Wound Drainage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Study knee related
Clicking/Popping/Crepitus/Grinding (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) — Study knee related
Pain (progressive/persistent) (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (10) — Study knee related
Baker's Cyst (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — Study knee related
Articular Surface Dislocation/Disassociation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Study knee related
Cellulitis/Redness/Blistering (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Study knee related
Effusion/Swelling/Edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) — Study knee related
Traumatic Injury (study knee) (Injury, poisoning and procedural complications) | 2 (3) | 3 (3) — Study knee related
Infection (not study knee) (Infections and infestations) | 3 (3) | 0 (0) — General adverse event (not study knee)
Other General Adverse Event (General disorders) | 4 (6) | 0 (0) — General adverse event (not study knee)
Musculoskeletal (not study knee)* (Musculoskeletal and connective tissue disorders) | 16 (24) | 12 (20) — General adverse event (not study knee)
Other Ipsilateral Knee Related Adverse Event (General disorders) | 2 (2) | 0 (0) — Study knee related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publication or presentation will be submitted to sponsor for review (not for approval or disapproval) at least thirty (30) days prior to submission for publication or presentation. If proposed publication or presentation contains patentable subject matter that needs protection, sponsor may request PI to delay the publication or presentation for an additional ninety (90) days to allow Sponsor to file a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT03272373/Prot_SAP_000.pdf